CLINICAL TRIAL: NCT02908906
Title: A First-in-Human, Open-label, Phase 1/2 Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of JNJ-63723283, an Anti-PD-1 Monoclonal Antibody, in Subjects With Advanced Cancers
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of JNJ-63723283, an Anti-PD-1 Monoclonal Antibody, in Participants With Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108223; 63723283LUC1001 (Other: Janssen Research & Development, LLC); 2016-002017-22 (EudraCT Number); 2023-506144-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- JNJ-63723283 (Experimental): In Part 1, the first cohort will receive JNJ-63723283 at a starting dose of 80 milligram (mg), intravenous (IV) every 2 weeks. JNJ-63723283 doses will be escalated following a modified Continual Reassessment Method (mCRM). Multiple doses, dose administration routes (subcutaneous [SC] or IV), and dose schedules may be explored. In Part 2, participants will receive JNJ-63723283 at the recommended Phase 2 dose (RP2D) determined in Part 1. In Part 3, participants will receive JNJ-63723283 to evaluate pharmacokinetic (PK), pharmacodynamic (PD) and safety. In Part 4, participants will receive JNJ-63723283 at the dose level determined in Part 3. Additional cohorts may be enrolled in Part 4.
  Interventions: Drug: JNJ-63723283

INTERVENTIONS:
Drug: JNJ-63723283 — JNJ-63723283 will be administered by IV infusion or SC injection or infusion.
  Other Names: Cetrelimab

SUMMARY:
The Primary purpose of this study is to identify the recommended Phase 2 dose [RP2D(s)] for JNJ-63723283 in Part 1, to assess the anti-tumor activity of JNJ-63723283 at the RP2D(s) in participants with selected advanced cancers including non-small-cell lung cancer (NSCLC), melanoma, renal, bladder, small-cell lung cancer (SCLC), gastric/esophageal cancer, and high-level microsatellite instability (MSI-H) or mismatch repair-deficient (dMMR) colorectal cancer (CRC) in Part 2, to determine one or more additional RP2Ds in Parts 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Parts 1-4: Have an Eastern Cooperative Oncology Group [ECOG] performance status 0 or 1
* Parts 1-4: Has thyroid function laboratory values within normal range
* Parts 1-4: Females of childbearing potential must have a negative serum pregnancy test
* Parts 1-4: Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* For Part 2 only: Participants enrolled into Part 2 must have tumor tissue available for correlative studies. Fresh tumor biopsy is preferred. Archival tissue must meet the following criteria: archival sections within 4 months of sectioning that have been stored at 2 degree to 8 degree Celsius in the dark or archival tumor blocks within 5 years of collection. Participants without tissues meeting the aforementioned archived tissue criteria must undergo a fresh biopsy
* Parts 1 to 4: Have evaluable disease

Exclusion Criteria:

* Has uncontrolled intercurrent illness, including but not limited to ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure (New York Heart Association class III-IV), unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension or diabetes, or psychiatric illness/social situation that would limited compliance with study requirements
* Has had prior treatment with an anti-Programmed-cell death receptor-1 (PD-1) antibody, anti-the ligand to programmed-cell death 1 (PD-L1) antibody or anti-the ligand to programmed-cell death 2 (PD-L2) antibody
* Treatment with any local or systemic anti-neoplastic therapy, radiotherapy (excluding limited palliative radiation), or investigational anticancer agent within 14 days or 4 half lives, whichever is longer, up to a maximum wash-out period of 28 days prior to the initiation of study drug administration
* Grade 3 or higher toxicity effects from previous treatment with immunotherapy
* A female who is pregnant, breast-feeding, or planning to become pregnant while enrolled in this study or within 5 months after the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Frequency and Severity of Dose-Limiting Toxicity (DLT) | Up to 2 years 6 months
  Frequency and severity of dose-limiting toxicity will be reported.
Part 2: Overall Response Rate (ORR) per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in Subjects With Selected Advanced Solid Tumors | Up to 2 years 6 months
  Objective Response Rate (ORR) is defined as percentage of subjects with best objective response of complete response (CR) or partial response (PR) based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) criteria.
Parts 3 and 4: Area Under the Serum Concentration Versus Time Curve from Time Zero to Dosing Interval (AUC [0-tau]) | Up to 2 years 6 months
  AUC (0-tau) is defined as area under the serum concentration versus time curve from time zero to dosing interval.

SECONDARY OUTCOMES:
Parts 1, 2, 3, and 4 : Number of Participants With Adverse Events (AEs) as a Measure of Safety | Up to 2 years 6 months
  An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment.
Parts 1, 2 and 3, and 4: Maximum Observed Serum Concentration (Cmax) | Up to 2 years 6 months
  The Cmax is the maximum observed serum concentration.
Parts 1 and 2: Area Under the Serum Concentration Versus Time Curve Between time t1 and t2 (AUC [t1-t2]) | Up to 2 years 6 months
  AUC (t1-t2) is defined as the area under the serum concentration versus time curve between time t1 and t2.
Parts 1, 2 and 3: Elimination Half-Life (t1/2) | Up to 2 years 6 months
  The elimination half-life (t1/2) is the time measured for the serum concentration to decrease by 1 half to its original concentration.
Parts 1 and 2: Total Systemic Clearance of (CL) | Up to 2 years 6 months
  Total systemic Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body.
Parts 1 and 2: Volume of Distribution at Steady-State (Vss) | Up to 2 years 6 months
  The Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of JNJ-63723283 at steady state.
Parts 1 and 2: Accumulation Ratio (R) | Up to 2 years 6 months
  The R is obtained by dividing AUC at two different time points.
Parts 3 and 4: Average Concentration (Cavg) of JNJ-63723283 | Up to 2 years 6 months
  Cavg of JNJ-63723283 will be reported.
Parts 3 and 4: Area Under the Serum Concentration Versus Time Curve Between Time Zero and Time t (AUC [0-t]) | Up to 2 years 6 months
  AUC (0-t) is defined as area under the serum concentration versus time curve between time zero and time t.
Parts 3: Area Under the Serum Concentration Versus Time Curve from Time Zero to Infinity (AUC [0-Infinity]) | Up to 2 years 6 months
  AUC (0-infinity) is defined as area under the serum concentration versus time curve from time zero to infinity.
Parts 3 and 4: Concentration Observed at the Last Timepoint Prior to Dosing (Ctrough) | Up to 2 years 6 months
  Ctrough is defined as the concentration observed at the last timepoint prior to dosing.
Parts 1, 2, 3, and 4: Presence of Anti-JNJ-63723283 Antibodies and Effect on Serum JNJ-63723283 Concentrations | Up to 2 years 6 months
  Serum samples will be analyzed for antibodies to JNJ-63723283. The titer of the confirmed positive samples will be reported.
Parts 1, 2, 3, and 4: Overall Response Rate (ORR) per Immune-Related Response Criteria (irRC) | Up to 2 years 6 months
  ORR is defined as percentage of subjects with best objective response of complete response (CR) or partial response (PR) based on irRC criteria.
Parts 1, 2, 3, and 4: Duration of Response (DOR) per RECIST v1.1 | Up to 2 years 6 months
  For Participants who achieve CR or PR, DOR will be calculated as time from initial response of CR or partial response (PR) to progressive disease or death due to underlying disease whichever comes first.
Parts 1, 2, 3, and 4: Duration of Response (DOR) per irRC | Up to 2 years 6 months
  For Participants who achieve CR or PR (defined by irRC), DOR will be calculated as time from initial response of CR or partial response (PR) to progressive disease or death due to underlying disease whichever comes first.
Parts 1, 2, 3, and 4: Clinical Benefit Rate (CBR) per RECIST v1.1 | Up to 2 years 6 months
  The CBR is defined as the percentage of participants who achieve CR, PR or stable disease (SD; greater than or equal to [>=] 24 weeks from the 1st study drug) based on RECIST v1.1 criteria.
Parts 1, 2, 3, and 4: Clinical Benefit Rate per irRC | Up to 2 years 6 months
  The CBR is defined as the percentage of participants who achieve CR, PR or SD (>= 24 weeks from the 1st study drug) based on irRC criteria.
Parts 1, 2, 3, and 4: Progression-free Survival (PFS) per RECIST v1.1 | Up to 2 years 6 months
  The time from first dose of JNJ-63723283 to progressive disease as defined by RECIST v 1.1 or death due to any cause.
Parts 1, 2, 3, and 4: Progression-free Survival (PFS) per irRC | Up to 2 years 6 months
  The time from first dose of JNJ-63723283 to progressive disease as defined by irRC or death due to any cause.
Parts 1, 2, 3, and 4: Overall Survival (OS) | Up to 2 years 6 months
  The time from first dose of JNJ-63723283 to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- United States (2):
  - St Louis, Missouri
  - Pittsburgh, Pennsylvania
- Chisinau, Moldova
- Poland (2):
  - Bialystok
  - Warsaw
- Russia (3):
  - Moscow
  - Pyatigorsk
  - Saint Petersburg
- Spain (7):
  - Badalona
  - Barcelona
  - Madrid
  - Málaga
  - Pamplona
  - Seville
  - Valencia
- Gothenburg, Sweden
- United Kingdom (4):
  - Glasgow
  - London
  - Manchester
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Felip E, Moreno V, Morgensztern D, Curigliano G, Rutkowski P, Trigo JM, Calvo A, Kowalski D, Cortinovis D, Plummer R, Maio M, Ascierto PA, Vladimirov VI, Cervantes A, Zudaire E, Hazra A, T'jollyn H, Bandyopadhyay N, Greger JG, Attiyeh E, Xie H, Calvo E. First-in-human, open-label, phase 1/2 study of the monoclonal antibody programmed cell death protein-1 (PD-1) inhibitor cetrelimab (JNJ-63723283) in patients with advanced cancers. Cancer Chemother Pharmacol. 2022 Apr;89(4):499-514. doi: 10.1007/s00280-022-04414-6. Epub 2022 Mar 17. PMID 35298698